CLINICAL TRIAL: NCT04889469
Title: Indications for Breast Reduction in the Public Health Care System
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-01508
Record Dates: First submitted 2021-04-24; First posted 2021-05-17 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Mammary Gland Hyperplasia
Keywords: breast reduction; reduction mammaplasty; breast hypertrophy
MeSH Terms: conditions — Gigantomastia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Breast hypertrophy operated: Women who have had a breast reduction in the public health care system
  Interventions: Procedure: Breast reduction
- Breast hypertrophy controls: Women with symptoms of breast hypertrophy, who do not fulfill the requirements to have a breast reduction in the public health care system
- Augmented controls: Patients who have breast hypertrophy due to cosmetic breast augmentation
- The general public: Random sample of the general public

INTERVENTIONS:
Procedure: Breast reduction — Procedure to remove excess fat, tissue and skin from the breasts.
  Groups: Breast hypertrophy operated

SUMMARY:
The overall purpose of the project is to create a scientific basis for which patients should be offered breast reduction in the public sector. More specifically , the project aims to:

* To examine the evidence for current national guidelines for breast reduction. The hypothesis is that BMI, breast volume, resection weight, and mental and physical symptoms affect the outcome of breast reconstruction, both in terms of complication risks, patient satisfaction and quality of life .
* To investigate which patients benefit the most from a breast reduction, in a health economic perspective. The starting point is that resources are limited and the purpose is to maximize the health effects for the patient at as low cost as possible. The hypothesis is that the health benefits, for the individual and society, are different depending on how big the breasts are and how much symptoms a patient has preoperatively.
* To examine back function and objective problems in women, with both natural and augmented breasts, with different body constitutions and volumes. The hypothesis is that a certain breast volume give rise to different physical symptoms in different women, depending on their other physical factors.
* To develop preferences for benign breast conditions that are treated in plastic surgery and for complications that the treatment can cause. Preferences are used to calculate QALY (quality-adjusted life years). Knowledge of preferences is essential for an analysis of healthcare needs.
* To examine women's experiences of how their breast hypertrophy affects them and their expectations of a breast reduction. The hypothesis is that the experience breast hypertrophy affects patients differently, and that expectations on a breast reduction can vary between different individuals.

ELIGIBILITY:
Inclusion Criteria:

* Breast volume > 800 ml
* BMI< 25 if under 50 years of age and BMI<2 if over the age of 50
* Symptoms of breast hypertrophy
* Non-smokers

Un-operad controls:

-Symptoms of breast hypertrophy, but do not comply with the criteria above.

Augmented controls:

* Augmented breast volume > 800 ml
* BMI< 25 if under 50 years of age and BMI<2 if over the age of 50

Exclusion Criteria:

* Inability to provide informed consent
* Inability to understand the Swedish language
* Age under 18 years

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Normal weight women with breast volumes over >800 ml (augmented or natural) with or without symptoms of breast hypertrophy. Normal weight women with a breast volume under 800 ml with symptoms of breast hypertrophy.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient reported quality of life | 5 years
  Breast -Q breast reduction preoperatively and postoperatively measures quality of life and patient satisfaction in 6 domains: physical well-being, psychosocial well-being, sexual well-being, satisfaction with the breasts, satisfaction with the result and satisfaction with care. Each domain is scored 0-100, where a higher score indicate a better outcome.
Complications | 1 year
  Complications after surgery classified according to Clavien-Dindo
Preferences (utility) | 5 years
  utility scores for various benign breast conditions that may require plastic surgery , including complications after cosmetic surgery, will be measured. Complications will be compared with situations without these , but also with congenital conditions that give a similar appearance. Measured with a visual analogue scale from 1-100.
Range of motion | 1 year
  Measured with goniometer in degrees
Muscle strength | 1 year
  Biering-Sörensen test measuring how many seconds the subject is able to keep the unsupported upper body horizontal, while placed prone with the buttocks and legs fixed to the couch by three wide canvas straps and the arms folded across the chest
Cost-effectiveness | 1 year
  Analysis of costs related to quality-adjusted life years, comparing operation with no operation.

SECONDARY OUTCOMES:
Patient reported health | 5 years
  EuroQol-5 dimensions - 3 levels -5D is a generic instrument developed for health economic and clinical evaluation of healthcare.A total score between 0 and 1 is calculated. = equals death and 1 perfect health.
Patient reported health | 5 years
  EQ VAS measures health on a scale from 0-100, where 100 equals perfect health and 0 worst possible health.
Body image | 5 years
  Multidimensional body-self relation questionnaire - appearance scales ( MBSRQ -AS).It is a 34-item self-report questionnaire designed to measure appearance related components of body-image. In consists of five subscales: appearance evaluation, appearance orientation, body areas satisfaction, overweight preoccupation, and self-classified weight. It is a 5-point Likert-scale ranging from 1 to 5.
Body investment | 5 years
  Appearance schemes inventory-revised ( ASI -R)is a 20-item self-report questionnaire designed to measure body-image investment. It consists of two subscales, self-evaluative salience (SES) and motivational salience (MS). It is a 5-point Likert-scale ranging from 1 (strongly disagree) to 5 (strongly agree). Twelve items relate to SES and eight items relate to MS. The total score is the mean of the 20 items, and the score of the subscales is the mean of the items relating to each subscale. A high score indicates greater body-image investment.
Pain intensity and quality | 5 years
  Short Form McGill Pain Questionnaire (SF- MPQ ).Measures pain on three subscales : a sensory subscale with 11 words, an affective subscale with 4 words that measures the quality of pain and a visual analogue scale (VAS) where the patient rates pain intensity from 1 to 10.
Pain intensity and effect on every-day life | 5 years
  Brief Pain Inventory -Short Form ( BPI -SF).Measures both pain intensity (sensory scale) and how pain affects the patient's life ( activity scale). The instrument also contains questions about pain relief, pain quality and the patient's experience of the cause of pain.The BPI scale defines pain as follows: Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Most important reason for operation | Pre-operative
  In-house designed questionnaire where patients preoperatively rank the most important reasons why they want to be operated on.
Most important effects of an operation | 1 year
  In-house designed questionnaire where patients postoperatively rank what the most important effects of the operation are.
The experience of breast hypertrophy and a breast reduction | 1 year
  The issues will be examined mainly with the help of semi-structured qualitative in-depth interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Hansson, PhD, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska university hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Widmark-Jensen E, Bernhardsson S, Eriksson M, Hallberg H, Jepsen C, Jivegard L, Liljegren A, Petzold M, Svensson M, Warnberg F, Hansson E. A systematic review and meta-analysis of risks and benefits with breast reduction in the public healthcare system: priorities for further research. BMC Surg. 2021 Sep 11;21(1):343. doi: 10.1186/s12893-021-01336-7. PMID 34511096
- See also: Health Technology Assessment (HTA) report 2021:121 — https://mellanarkiv-offentlig.vgregion.se/alfresco/s/archive/stream/public/v1/source/available/sofia/su4372-1728378332-394/native/2021_121%20HTA-rapport%20Bröstreduktion.pdf